CLINICAL TRIAL: NCT07337083
Title: Screening of Prediabetes in End Stage Renal Disease on Dialysis
Brief Title: Prediabetes in End Stage Renal Disease on Dialysis
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hany Ahmed Mohamed, lecturer of internal medicine, Sohag University
Other Study IDs: Soh-Med-25-4--6PD
Record Dates: First submitted 2026-01-04; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-04

CONDITIONS: Screening; Pre Diabetic; Chronic Renal Failure (CRF); Dialysis Patients
MeSH Terms: conditions — Glucose Intolerance; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prediabetes is a highly prevalent condition, affecting about one-third of adults in the United States Patients with prediabetes have an increased risk for diabetes, with 2% to 10% progressing to diabetes each yea Although prediabetes is frequently considered an intermediary stage in the progression between normoglycemia and diabetes, many individuals may have prediabetes for several years, while some may never progress.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease on dialysis patients aged ≥ 18 years old.

Exclusion Criteria:

1. Patients previously diagnosed with prediabetes.
2. Patients previously diagnosed with diabetes mellitus.
3. Acute Medical Status :Hospitalized patients.
4. Physiological States: Pregnant females.Lactating females.
5. Specific Comorbidities & Conditions: Polycystic kidney disease.
6. New York Heart Association (NYHA) class III or IV heart failure.
7. Known liver cirrhosis. or HIV/AIDS.
8. Renal cancer.
9. Active immunosuppression. or Recent chemotherapy or immunosuppressive therapy.
10. History of organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is defined as adult patients (aged 18 years or older) with End-Stage Renal Disease (ESRD) who are currently on dialysis.
  This population will be recruited from a single center: Sohag Faculty of Medicine, Sohag University, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2025-04-13 (Actual); Primary Completion 2025-09-13 (Actual); Study Completion 2025-10-12 (Actual)

PRIMARY OUTCOMES:
The prevalence of prediabetes in the End Stage Renal Disease (ESRD) on dialysis cohort. | "The time frame for measurement of the primary outcome (prevalence of prediabetes) with all diagnostic measurements (Fasting Plasma Glucose mg/dl) performed once per participant at the time of their inclusion in the study."

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Sohag, Egypt
  - Sohag University .Faculty of Medicine, Sohag

IPD SHARING:
Plan to Share IPD: Undecided